CLINICAL TRIAL: NCT01321593
Title: Comparison of the Hemoglobin Results Obtained With the "Orsense NBM-200MP" Device and the Clinical Laboratory
Brief Title: Hemoglobin Measured by "Orsense NBM-200MP" Device and Laboratory Measurement
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/28; 2010-A00541-38 (Other: ANSM)
Record Dates: First submitted 2011-03-19; First posted 2011-03-23 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hemoglobin determination: emergency unit patients

SUMMARY:
The purpose of this study is to compare the hemoglobin results obtained with the "Orsense NBM-200MP" device and the Clinical Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* emergency unit patients requiring an hemoglobin determination

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency unit patients requiring an hemoglobin determination
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin measurement using the "Orsense NBM-200MP" device | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

REFERENCES:
- [Derived] Gayat E, Aulagnier J, Matthieu E, Boisson M, Fischler M. Non-invasive measurement of hemoglobin: assessment of two different point-of-care technologies. PLoS One. 2012;7(1):e30065. doi: 10.1371/journal.pone.0030065. Epub 2012 Jan 6. PMID 22238693